CLINICAL TRIAL: NCT06164522
Title: Prediction of Intraoperative Adhesions Before Cesarean Section: Integrating Parameters From History, Examination, and Investigations
Brief Title: Prediction of Intraoperative Adhesions Before CS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Ahmed Essa, Doctor, Assiut University
Other Study IDs: Intraoperative adhesions
Record Dates: First submitted 2023-12-02; First posted 2023-12-11 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Abdominal Adhesion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Abdominal ultrasound — Abdominal ultrasound to detect sliding sign

SUMMARY:
To predict the presence of intra-abdominal adhesions among women undergoing repeated cesarean section using several parameters.

DETAILED DESCRIPTION:
One of the most frequently performed surgical procedures globally is cesarean delivery (CD). Cesarean delivery rate is increasing, which raises the prevalence of intra-abdominal adhesions . The rate of intra-abdominal adhesions is 24-83% . Adhesions cause various postoperative complications, including intestinal obstruction, pelvic pain, dyspareunia, infertility, visceral injury, delayed delivery of the newborn , prolong surgical duration, increase bleeding amount and the incidence of hysterectomy . For these reasons, obstetricians always want to identify the possible extent of adhesions before cesarean section. Although to date there was no reliable technique to predict adhesions in women undergoing repeat CD .

Methods used in the evaluation of adhesions include the previous cesarean scar features, pigmentation, width and length , ultrasound sliding sign has been used in predicting pelvic endometriosis ,Baron et al. ,used the sliding sign in predicting adhesions in women undergoing repeat CD, also Stretch marks are a type of skin alteration that occur during pregnancy.

To ensure better surgical outcomes and reduce morbidities, the accurate prediction of adhesion formations before cesarean section is important. This study aims to investigate the integration of multiple parameters, such as evaluating cesarean scars, ultrasound sliding sign, and striae gravidarum, to assess intra-abdominal adhesions. We hypothesize that employing a combination of these parameters will yield superior predictive capabilities compared to relying on a single parameter alone. By exploring a comprehensive approach to adhesion prediction, we endeavor to enhance the safety and efficacy of cesarean section procedures, ultimately improving maternal and fetal well-being.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women aged from 18 to 35 years
2. Women with at least one previous C-section
3. Gestational age (≥36 weeks)
4. Planned elective cesarean section

Exclusion Criteria:

1. primigravida
2. Gestational age (<36 weeks)
3. Pregnant woman who had developed wound site infections following prior cesarean section

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: 1. Pregnant women aged from 18 to 35 years
  2. Women with at least one previous C-section
  3. Gestational age (≥36 weeks)
  4. Planned elective cesarean section
Sampling Method: Non-Probability Sample
Enrollment: 146 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Predicting presence of intra-abdominal adhesions among women undergoing repeated cesarean section using several parameters. | From January 2024 to February 2025
  Detection of intra-operative adhesions before repeated cesarean section by history, examination and ultrasound

REFERENCES:
- [Background] Shenhav S, Grin L, Kapustian V, Anteby EY, Gdalevich M, Gemer O. Quantifying the effects of postcesarean adhesions on incision to delivery time. J Matern Fetal Neonatal Med. 2019 Aug;32(15):2500-2505. doi: 10.1080/14767058.2018.1439010. Epub 2018 Feb 20. PMID 29415600
- [Background] Mokhtari M, Yaghmaei M, Akbari Jami N, Roudbari M, Jalalvand D. Prediction of Intraperitoneal Adhesions in Repeated Cesarean Section Using Sliding Sign, Striae Gravidarum, and Cesarean Scar. Med J Islam Repub Iran. 2022 May 2;36:44. doi: 10.47176/mjiri.36.44. eCollection 2022. PMID 36128300
- [Background] Piessens S, Edwards A. Sonographic Evaluation for Endometriosis in Routine Pelvic Ultrasound. J Minim Invasive Gynecol. 2020 Feb;27(2):265-266. doi: 10.1016/j.jmig.2019.08.027. Epub 2019 Sep 4. PMID 31493569
- [Background] Awonuga AO, Fletcher NM, Saed GM, Diamond MP. Postoperative adhesion development following cesarean and open intra-abdominal gynecological operations: a review. Reprod Sci. 2011 Dec;18(12):1166-85. doi: 10.1177/1933719111414206. Epub 2011 Jul 20. PMID 21775773
- [Background] Dogan NU, Haktankacmaz SA, Dogan S, Ozkan O, Celik H, Eryilmaz OG, Doganay M, Gulerman C. A reliable way to predict intraabdominal adhesions at repeat cesarean delivery: scar characteristics. Acta Obstet Gynecol Scand. 2011 May;90(5):531-4. doi: 10.1111/j.1600-0412.2011.01080.x. Epub 2011 Mar 16. PMID 21306338